CLINICAL TRIAL: NCT05275556
Title: Gastroenterology Artificial INtelligence System for Detecting Colorectal Polyps (The GAIN Study)
Acronym: GAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 103820
Record Dates: First submitted 2022-02-25; First posted 2022-03-11 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2023-12

CONDITIONS: Colon Adenoma; Colon Polyp; Colon Lesion
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Subjects, investigators, study site personnel, and pathologists will not be blinded to treatment assignments. All Verily personnel involved in the statistical analysis of this study will be blinded to treatment assignment. For the interim analysis, unblinded analysis will be performed by an independent statistician, the results of which will be communicated to a select group of Verily personnel not involved in the study management.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Colonoscopy (Standard of Care) (No Intervention): The control arm is colonoscopy with High Definition White Light Endoscopy (HD-WLE) per standard of care.
- CADe Device (Experimental): The intervention arm is colonoscopy with HD-WLE per standard of care plus the CADe Device.
  Interventions: Device: Computer-Assisted Detection (CADe) Device

INTERVENTIONS:
Device: Computer-Assisted Detection (CADe) Device — The CADe Device uses artificial intelligence to aid in identifying colorectal polyps during High Definition White Light Endoscopy (HD-WLE) based colonoscopies. This device connects the Gastroenterologist's colonoscopy video output source to the main monitor and highlights the regions of interest where the device detects a potential lesion. The CADe Device overlays graphical markers onto video from the endoscope camera and does not perform further processing to the endoscope video signal. This device is not intended to replace clinical decision making.
  Arms: CADe Device

SUMMARY:
This is a prospective, multicenter, randomized controlled study to evaluate the effect of the Computer-Assisted Detection (CADe) Device on Adenomas Per Colonoscopy and Positive Percent Agreement for routine colonoscopies. The control arm is colonoscopy performed with High Definition White Light Endoscopy (HD-WLE) per standard of care. The intervention arm is colonoscopy performed with HD-WLE per standard of care plus the Computer-Assisted Detection (CADe) Device.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo routine screening (including, but not limited to, FIT/Cologuard positive), routine surveillance (≥3 years as scheduled since last colonoscopy), or diagnostic (symptomatic) colonoscopy with High Definition White Light Endoscopy.
* Between the ages of 45 and 80 years, inclusive
* Able and willing to provide written informed consent

Exclusion Criteria:

* Self-reported pregnancy
* Known diagnosis of Colorectal Cancer
* History of, or referral for, Inflammatory Bowel Disease
* Previous surgery involving the colon or rectum
* Referral for known polyp or assessment of post-polypectomy site (i.e. less than 3 years since last colonoscopy).
* High suspicion or diagnosis of genetic polyposis syndromes, including familial adenomatous polyposis (FAP), hereditary nonpolyposis colorectal cancer (HNPCC), or any other high-risk family history meeting Bethesda guidelines.
* Referral for overt, symptomatic gastrointestinal bleeding

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scooter Plowman, MD, Study Director — Verily Life Sciences LLC
Locations (7):
- United States (5):
  - Mayo Clinic, Rochester, Minnesota
  - Duke Health, Durham, North Carolina
  - Great Lakes Gastroenterology Research, Mentor, Ohio
  - Susquehanna Research Group, Camp Hill, Pennsylvania
  - ANRC Research, El Paso, Texas
- Israel (2):
  - Elisha Medical Center, Haifa
  - Sourasky Medical Center (Ichilov), Tel Aviv

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Started | 694 | 716
Completed | 694 | 713
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colonoscopy (Standard of Care) | CADe Device | Total
Number analyzed (Participants) | 694 | 713 | 1407
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.42 (8.94) | 60.66 (9.16) | 60.54 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 369 | 383 | 752
  Male | 325 | 330 | 655
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 5
  Black or African American | 22 | 26 | 48
  White | 652 | 666 | 1318
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United States | 551 | 561 | 1112
  Israel | 143 | 152 | 295
Colonoscopy Indication [Count of Participants; unit: Participants]
  Screening | 373 | 377 | 750
  Surveillance | 277 | 281 | 558
  Diagnostic (symptomatic) | 44 | 55 | 99

OUTCOME MEASURES:

1. Primary Outcome: Difference in Adenomas Per Colonoscopy (APC)
Description: Difference in Adenomas Per Colonoscopy (APC) between the control and intervention arm, evaluated for superiority. APC is defined as the average number of histologically confirmed adenomas resected per colonoscopy.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Resected adenomas
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Resected adenomas | 0.60 [0.56 to 0.64] | 0.74 [0.71 to 0.77]
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Superiority; p = 0.0002, Poisson Regression — Threshold for significance is 0.025; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.07 to 0.23]

2. Primary Outcome: Difference in Positive Percent Agreement (PPA)
Description: Difference in Positive Percent Agreement (PPA) between the control and intervention arm, evaluated for non-inferiority. PPA is defined as the total number of histologically confirmed Clinically Significant Excised Lesions, divided by the total number of excisions.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of significant lesions
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Proportion of significant lesions | 0.62 [0.58 to 0.66] | 0.56 [0.52 to 0.60]
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Non-Inferiority — Non-inferiority margin is -10%; p = 0.09, Resampling based — Threshold for significance is 0.025; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.15 to 0.03]

3. Secondary Outcome: Adenoma Detection Rate (ADR)
Description: The Adenoma Detection Rate is defined as the number of patients with at least one histologically confirmed adenoma divided by the total number of patients enrolled per study arm.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Number (95% Confidence Interval); unit: Percentage of participants with adenomas
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Percentage of participants with adenomas | 38.9 [35.3 to 42.6] | 42.9 [39.2 to 46.6]
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Superiority; p = 0.031, Cochran-Mantel-Haenszel; Threshold for significance is 0.025; Difference in percentage = 5.5, 95% CI 2-sided [-0.3 to 11.2]

4. Secondary Outcome: Number of False Alerts Per Procedure
Description: A false alert is defined as a bounding box that persists on the screen (approximately 2-3 seconds per the judgment of the colonoscopist) that is then determined by the colonoscopist not to contain a polyp. The false alert rate is calculated as the number of false alerts per procedure conducted in the intervention arm of the study.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Number; unit: Number of false alerts
Arm/Group | CADe Device
Number analyzed (Participants) | 713
Number of false alerts | 417
Statistical Analysis 1: Comparison: CADe Device; Test type: Other; rate = 0.58

5. Secondary Outcome: Mean Withdrawal and Inspection Time (MWT)
Description: The withdrawal time is defined as the time measured from the moment the withdrawal phase of the procedure begins (with the scope in the cecum) to the moment the scope is withdrawn from the patient. The Inspection time measurement will exclude washing and resection, and other peri-resection activity not deemed to be colonic inspection. Inspection times for both the control arm and intervention arm will be calculated retrospectively upon review of the video recordings.
Time Frame: Day 1
Population: Convenience sample of available videos
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 660 | 669
minutes | 8.97 (4.97) | 9.34 (4.08)
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Other — 2 sided test for differences between arms; p = 0.169, Permutation test; Mean Difference (Final Values) = 0.58

6. Secondary Outcome: Polyp Detection Rate (PDR)
Description: Polyp detection rate is defined as the proportion of patients with at least one histologically-confirmed polyp detected.
Time Frame: Day 1
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 364 | 425
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Other; Descriptive analysis: 52.4 in Colonoscopy (Standard of Care), 59.6 in CAD-e Device

7. Secondary Outcome: Proximal Adenoma Detection Rate (pADR)
Description: pADR is defined as the percentage of patients with at least one histologically-confirmed adenoma detected in proximal colon.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 198 | 236
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Difference in percentage between both arms is reported. H0: Colonoscopy (Standard of Care) percentage <= CADe Device percentage (i.e. test of superiority); Test type: Superiority; p = 0.0578, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Net) = 4.6, 95% CI 2-sided [-0.2 to 9.4]

8. Secondary Outcome: Flat Adenoma Detection Rate (fADR)
Description: fADR is defined as the percentage of patients with at least one histologically-confirmed non-polypoid adenoma detected.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 19 | 21
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.7813, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.5 to 2.0]

9. Secondary Outcome: Serrated Lesions Per Colonoscopy (SLPC)
Description: SLPC is defined as the number of histologically confirmed serrated lesions detected, divided by the total number of colonoscopies.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: serated lesions per colonoscopy
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
serated lesions per colonoscopy | 0.34 [0.30 to 0.38] | 0.46 [0.42 to 0.50]
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Superiority; Least-squares means = 0.11, 95% CI 2-sided [0.05 to 0.17]

10. Secondary Outcome: Serrated Lesions Detection Rate (SLDR)
Description: SLDR is defined as the percentage of patients with at least one histologically confirmed serrated lesion detected.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 156 | 219
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [3.7 to 12.9]

11. Secondary Outcome: Adenoma Detection Rate Including Carcinoma (ADR*)
Description: ADR* is defined as ADR, but also includes histologically-confirmed intramucosal carcinoma and adenocarcinoma.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 271 | 307
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.1185, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-1 to 9.1]

12. Secondary Outcome: Small Adenoma Detection Rate (sADR)
Description: sADR is defined as the percentage of patients with at least one adenoma 5mm or smaller detected.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 201 | 236
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0752, Cochran-Mantel-Haenszel — nominal p-value; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [-0.4 to 9.2]

13. Secondary Outcome: Polyps Per Colonoscopy (PPC)
Description: PPC is defined as the total number of histologically-confirmed polyps found divided by the total number of colonoscopies performed, per study arm.
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Polyps per colonoscopy
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Polyps per colonoscopy | 1.03 [0.95 to 1.11] | 1.32 [1.24 to 1.41]

14. Secondary Outcome: Advanced Adenoma Detection Rate (aADR)
Description: aADR is defined as the percentage of patients with at least one adenoma ≥ 10 mm, or any adenoma < 10 mm, which was either of high-grade dysplasia (HGD) or villous or tubulovillous.
Time Frame: Day 1
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Participants | 60 | 59
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.8194, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.2 to 2.6]

15. Secondary Outcome: False Positive Rate (FPR)
Description: FPR is defined as the proportion of colorectal lesions resected and biopsied and subsequently not histologically-confirmed to be clinically relevant colorectal polyps (e.g. a pathology finding of normal mucosa, inflammatory tissue, stool or debris, lymphoid aggregates).
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of resected lesions
Units Other Than Participants: Resected lesions
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
Number analyzed (Participants) | 694 | 713
Number analyzed (Resected lesions) | 715 | 939
proportion of resected lesions | 0.22 [0.19 to 0.26] | 0.31 [0.28 to 0.35]
Statistical Analysis 1: Comparison: Colonoscopy (Standard of Care) vs CADe Device; Test type: Other — Test for difference; p = 0.0008, Exact poisson — Nominal p-value; Incidence Rate Ratio = 1.39, 95% CI 2-sided [1.14 to 1.69]

ADVERSE EVENTS:
Time Frame: 1 day
Description: An AE is defined as any untoward medical occurrence, unintended disease or injury in subjects, users or other persons, that is considered a change from baseline or pre-study status, whether or not related to the investigational medical device. Any pre-existing medical condition or symptoms present in a subject will not be considered an AE in this study, unless it worsens as a result of this study. For this study, AEs related to the study device and study procedures will be reported.
Arm/Group | Colonoscopy (Standard of Care) | CADe Device
All-Cause Mortality (participants affected / at risk) | 0/694 | 0/713
Serious Adverse Events (participants affected / at risk) | 0/694 | 0/713
Other Adverse Events (participants affected / at risk) | 0/694 | 0/713

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish, but there are limitations to protect confidential information and/or allow the sponsor to publish first.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT05275556/Prot_SAP_000.pdf